CLINICAL TRIAL: NCT03543982
Title: An Open-label, Pilot Study to Assess the Effects of an Oral Probiotic Product on the Vaginal Microbial Community and on Parameters of Vaginal Health
Brief Title: Effects of Oral Probiotic Product on Vaginal Microbial Community and Parameters of Vaginal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UAS Labs LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAS1RPD-160001-PRVH
Record Dates: First submitted 2018-04-27; First posted 2018-06-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Vaginal Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral probiotic product (Experimental)
  Interventions: Dietary Supplement: Oral probiotic product

INTERVENTIONS:
Dietary Supplement: Oral probiotic product — Once per day (QD), 28 days

SUMMARY:
The purpose of the study is to assess the efficacy and safety of an oral probiotic product on the vaginal microbiome and on parameters of vaginal health. Eligible subjects will utilize the investigational product as directed for a period of 28 days. The vaginal microbial community and parameters of vaginal health will be measured at baseline and after 14 and 28 days of supplementation. A follow-up post-supplementation visit will be conducted on Day 42.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women aged 18-50 years.
2. Body mass index 18.5 - 34.9 kg/m2 (inclusive).
3. Have childbearing potential [i.e. not surgically sterile or post-menopausal (greater than one year since last menses)].
4. Non-smoker, or ex-smoker ≥6 months.
5. Nugent score of 4-6 or pH >4.5
6. Agrees to maintain current level of physical activity and dietary habits throughout the trial period.
7. Agrees to discontinue use of probiotic supplements (oral or vaginal), as well as food supplemented with probiotics or prebiotics.
8. Willing and able to provide written informed consent.
9. Agrees to provide fecal samples during the trial period.

Exclusion Criteria:

1. Hypersensitivity to any ingredient in the study product.
2. Pregnancy or planning pregnancy.
3. Lactation or breast feeding.
4. Irregular menstrual cycles.
5. Use of contraceptives that contain spermicidal agents.
6. Use of an intrauterine device (IUD).
7. Use of hormonal therapy through cervical cap.
8. Use of douching devices.
9. Any major trauma or surgical event within the 3 months prior to screening.
10. Individuals undergoing therapies to prevent any recurrent infections.
11. Allergy to any antibiotic that may be prescribed as a rescue remedy during the study.
12. Use of prescription drugs (other than birth control) within 1 month prior to Visit 1.
13. Use of antibiotics within 2 months prior to Visit 1.
14. History of blood clotting disorders or use of coagulation-inhibiting drugs (e.g. warfarin)
15. Presence of systemic diseases or immunodeficiencies
16. Abdominal or gastrointestinal surgery within the previous 12 months.
17. Recent gastrointestinal food-borne illness (within 1 month prior to Visit 1)
18. History of cancer (excluding non-melanoma skin cancer and basal cell carcinoma) in the past 5 years
19. Abnormal laboratory test results of clinical significance
20. Presence or history (past 6 months) of alcohol or drug abuse
21. Subject is unwilling or unable to abide by the requirements of the protocol
22. Any condition that would interfere with the subject's ability to comply with study instructions, might confound the interpretation of the study, or put the subject at risk
23. Subject has taken an investigational health product or has participated in a research study within 30 days prior to first study visit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Changes in vaginal microbial community, via next generation sequencing. | Day 28

SECONDARY OUTCOMES:
Changes in vaginal microbial community, via next generation sequencing. | Day 14 and 42
Changes in vaginal pH. | Day 14, 28 and 42
Changes in Nugent Score (Scale of 0 to 10). | Day 14, 28 and 42
Parameters of well-being, via Vulvovaginal Symptom Questionnaire. | Day 14, 28 and 42
Safety as assessed by routine chemistry and hematology, and the monitoring of adverse events. | Day 14, 28 and 42
Compliance as assessed by capsule counts of the returned IP. | Day 14, 28 and 42

OTHER OUTCOMES:
Colonization of the vaginal microbiome. | Day 14, 28 and 42
Colonization of the GI microbiome. | Day 14, 28 and 42

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrasource, Guelph, Ontario, Canada